CLINICAL TRIAL: NCT05565781
Title: Impact of Non-invasive Remote Monitoring Via Wearable Technologies for Detection of Atrial Fibrillation in Patients With Cryptogenic Stroke
Brief Title: Smartwatch and External Holter Monitoring to Detect Atrial Fibrillation in Patients With Cryptogenic Stroke
Acronym: SMARTTHUNDER
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Universitari Vall d'Hebron Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: PI20/01210
Record Dates: First submitted 2022-09-21; First posted 2022-10-04 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-04

CONDITIONS: Paroxysmal Atrial Fibrillation; Cryptogenic Stroke
Keywords: Wearable Electronic Devices
MeSH Terms: conditions — Atrial Fibrillation; Ischemic Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- ECG Smartwatch for up to 1 year (Active Comparator): Cardiac monitoring with a smartwatch that support the recording of a single-lead electrocardiogram (ECG) over 1 year after the acute phase of cryptogenic stroke. Simultaneously, a continuous cardiac monitoring will be performed using an Insertable Cardiac Monitor (ICM)
  Interventions: Device: ECG smartwatch; Device: Insertable Cardiac Monitor (ICM)
- Holter monitoring for up to 1 year (Active Comparator): Cardiac monitoring with an external holter device for 30 days after the acute phase of cryptogenic stroke and 15 additional days of extended use every 3 months up to 1 year
  Interventions: Device: External ECG Monitoring
- Control group (Other): Regular cardiac monitoring with an external holter device for 30 days after the acute phase of cryptogenic stroke
  Interventions: Device: External ECG Monitoring

INTERVENTIONS:
Device: ECG smartwatch — Testing ECG smartwatch to detect AF or potential signs of AF
  Arms: ECG Smartwatch for up to 1 year
Device: Insertable Cardiac Monitor (ICM) — Gold-standard cardiac monitor for comparison of testing device (ECG smartwatch)
  Arms: ECG Smartwatch for up to 1 year
Device: External ECG Monitoring — Regular cardiac monitor for diagnosis of AF
  Arms: Control group; Holter monitoring for up to 1 year

SUMMARY:
Stroke recurrence largely depends on the detection of the cause and the control of vascular risk factors, with occult atrial fibrillation (AF) being one of the most important. Prolonged ambulatory cardiac monitoring is recommended for detecting occult AF. Currently, there are non-invasive monitoring devices such as the textile Holter that have proven to be useful for monitoring for up to 30 days but not longer. Another alternative is smartwatches, although they must be validated for use in the elderly population who have had a stroke.

DETAILED DESCRIPTION:
The primary objective is to demonstrate that the protocol of ambulatory cardiac monitoring with wearable devices for 12 months allows detection of a higher percentage of occult AF than monitoring for 30 days. The secondary objectives will be to demonstrate the internal validity of smartwatches against insertable cardiac recorders for the detection of AF. To evaluate the usability and adherence to the use of smartwatches in patients with stroke. Detect predictors that can help detect long-term occult AF. Determine the profile of vascular events in each group. Detect predictors of vascular recurrence defined as stroke recurrence, incidence of cerebral hemorrhage, heart failure, myocardial infarction or vascular death.

ELIGIBILITY:
Inclusion Criteria:

* Age greater to or equal to 55 years
* Patients with diagnosis of cryptogenic stroke after a basic study that included neuroimaging, extra/intracranial vascular evaluation, 24-hour monitoring, and echocardiogram
* Patients with acute cortical infarction with the presence of intracranial occlusion (preferably)
* Modified Rankin Scale (mRS) lower to 4

Exclusion Criteria:

* Diagnosis of lacunar infarction or transient ischemic attack (TIA)
* Diagnosis of stroke of known source: atherothrombotic due to moderate or severe symptomatic extra/intracranial stenosis, major cardioembolic cause (atrial fibrillation, anterior or apical ventricular akinesis, causal PFO, post-AMI, flutter or mitral stenosis), unusual cause (thrombophilia, arterial dissection symptomatic, toxic)
* Use of pacemakers
* Circumstances that may preclude the clinical follow-up or reduce the possibilities of obtaining data to achieve the objectives of the study and/or limit contact with the investigator (for example, transfer to a social health center)
* Unwillingness to the use of cardiac monitoring wearable devices
* Not understanding study procedures

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-03-28 (Actual); Primary Completion 2025-06-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Increased probability of detecting AF | Assessed throughout 1 year trial period
  To identify and compare prevalence rates of AF detection for the purpose of determine the clinical relevance or not of a prolonged screening process for AF. On the intervention group, patients will have a cardiac monitoring for up to 12 months. If AF is detected by ECG smartwatch, the ICM data will be analyzed by a cardiologist team and provide an ECG report to investigators in order to confirmed ECG smartwatch result.

SECONDARY OUTCOMES:
Identification of Atrial Fibrillation using a ECG smartwatch | Assessed throughout 1 year trial period
  Episodes of atrial fibrillation detected by the ECG smartwatch will be compared to the gold-standard cardiac monitor
Usability and adherence to ECG Smartwatch | Assessed throughout 1 year trial period
  To evaluate the usability to the use of the ECG Smartwatch through the System usability scale (SUS) and self-reported of likes or dislikes encountered with wearable.
Control of vascular risk factors (VRF) | Assessed at the end of the 1 and 2 year trial period
  To describe and compare the percentage of adequate control of VRFs among patients in each study group. VRFs metrics are defined according to the American Heart Association's recommendations, including blood pressure, lipids, glucose, body mass index, nicotine exposure, diet, physical activity, and sleep health. Sub-study analysis will be perform considering data from smartwatch such as sleep, physical activity, and other health behavior.
Vascular events incidence | Assessed at the end of the 1 and 2 year trial period
  To describe the vascular events defined as recurrence of stroke, the incidence of cerebral hemorrhage, heart failure, myocardial infarction, or vascular death in each study group
Predictors of vascular recurrence | Assessed at the end of the 1 and 2 year trial period
  To identify predictors of vascular recurrence (recurrent stroke, cerebral hemorrhage, heart failure, myocardial infarction, or vascular death) in each study group. Predictors of vascular recurrence included sociodemographic data such as age, sex and education level; BMI (kg/m2); history of diabetes mellitus; LDL-cholesterol and medications, such as the use of anti-hypertensive medications, lipid-lowering medications, and antiplatelet therapy. Also clinical symptoms, neuroimagen and ECG parameters will be included in the analysis.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitari Vall d'Hebron, Barcelona, Catalonia, Spain

IPD SHARING:
Plan to Share IPD: No